CLINICAL TRIAL: NCT05012111
Title: The Natural History of Acquired and Inherited Bone Marrow Failure Syndromes
Brief Title: Natural History of Acquired and Inherited Bone Marrow Failure Syndromes
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000387; 000387-H
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01-16

CONDITIONS: Severe Aplastic Anemia; Telomere Biology Disorders; Inherited Bone Marrow Failure Syndromes
Keywords: Aplastic Anemia; Telomere; Natural History
MeSH Terms: conditions — Anemia, Aplastic; Congenital Bone Marrow Failure Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Severe Aplastic Anemia(SAA): Age 2 and older; Previous diagnosis of bone marrow failure
- Cohort 2: Other Marrow Failure: Age 2 and older; Previous diagnosis of bone marrow failure;
- Cohort 3: Telomere Biology Disorders(TBD): Age 2 and older; Previous diagnosis of bone marrow failure
- Cohort 4: Inherited Bone Marrow Failure(IBMF)Syndromes: Age 2 and older; Previous diagnosis of bone marrow failure
- Cohort 5: Family Screening: Age 2 and older; First degree family member with a known or suspected inherited bone marrow failure syndrome

SUMMARY:
Background:

Bone marrow failure diseases are rare. Much is known about the diseases at the time of diagnosis, but long-term data about the effects of the diseases and treatments are lacking. Researchers want to better understand long-term outcomes in people with these diseases.

Objective:

To follow people diagnosed with acquired or inherited bone marrow failure disease and study the long-term effects of the disease and its treatments on organ function.

Eligibility:

People aged 2 years and older who have been diagnosed with acquired or inherited bone marrow failure or Telomere Biology Disorder. First degree family members may also be able to take part in the study.

Design:

Participants will be screened with a medical history, physical exam, and blood tests. They may have a bone marrow biopsy and aspiration. For this, a large needle will be inserted in the hip through a small cut. Marrow will be drawn from the bone. A small piece of bone may be removed.

Participants may also be screened with some of the following:

Cheek swab or hair follicle sample

Skin biopsy

Urine or saliva sample

Evaluation by disease specialists (e.g., lung, liver, heart)

Imaging scan of the chest

Liver ultrasounds

Six-Minute Walk Test

Lung function test

Participants will be put into groups based on their disease. They will have visits every 1 to 3 years. At visits, they may repeat some screening tests. They may fill out yearly surveys about their medicines, transfusions, pregnancy, bleeding, and so on. They may have other specialized procedures, such as imaging scans and ultrasounds.

Participation will last for up to 20 years.

DETAILED DESCRIPTION:
Study Description: This study will allow for the long term follow up of patients with acquired and inherited bone marrow failure, both treated and untreated.

Objectives:

Primary Objective

The primary objective is to characterize disease and treatment related long-term outcomes in subjects with inherited or acquired marrow failure.

Secondary Objectives

1. Rates of disease progression requiring intervention
2. Determine overall survival
3. Determine event free survival in subjects who receive treatment
4. Genetic or molecular biomarker to predict the long-term outcomes/early diagnosis in SAA and disease progression in other marrow failures.
5. Determine effects of pregnancy, viral infections, and vaccinations on disease course
6. Determine rates of both hematologic and solid organ malignancies
7. For Telomere Biology Disorders (TBD) cohort, assess the systemic impact of the disease including lung function, liver function, immunodeficiency, endocrine disorders, vascular disorders, and cardiovascular disease
8. For diseases with a genetic cause, determine the differences in clinical phenotype between different mutations causing the syndrome (example within TBD)
9. Family genetic studies to determine the incidence and penetrance of specific gene mutations within one family

Tertiary/Exploratory Objectives

1. Genomic analysis (including whole exome or whole genome sequencing) to seek a potentially disease-causing mutations in subjects who meet the clinical phenotype for inherited disease but do not harbor a known mutation using sequencing
2. Serial assessment of hematopoiesis and immune activity as it relates to clinical course

Endpoints:

Primary Endpoints:

Cohort 1 (SAA): Rate of relapse and clonal evolution in previously treated subjects.

Cohort 2 (Other Marrow Failure): Rate of progression (cytopenias or clonal evolution) requiring therapeutic intervention.

Cohort 3 Telomere Biology Disorders (TBD): Development of cytopenias, lung disease or liver disease, or (if present at baseline)

characterization, and rate of progression of cytopenias, lung disease or liver disease in TBD subjects and looking at their overall contribution to morbidity and mortality.

Cohort 4 Inherited Bone Marrow Failure (IBMF): Rate of progression to transfusion dependent marrow failure, marrow failure requiring therapeutic intervention (such as medical therapy or HSCT) or the progression to hematological or solid malignancy.

Secondary Endpoints:

Cohort 1 (SAA):

1. Response to treatment at 3 and 6 months and rates of relapse
2. Overall survival
3. Type and severity of additional medical diagnoses
4. Rates of clinically significant paroxysmal nocturnal hemoglobinuria (PNH)
5. Rates, timing, and treatment of abnormal iron status (iron overload or deficiency)
6. Rates and outcomes of pregnancy, and rate and treatment of abnormal menses
7. Rates of drug induced complications
8. Incidence of vaccination and rates of relapse following administration

Cohort 2 (Other Marrow Failure):

1. Treatment response
2. Development of PNH and occurrence of symptoms, or need for therapy
3. Overall survival

Cohort 3 (TBD):

1. Overall survival
2. Response to treatment in terms of improvement of cytopenias, or slower progression of lung or liver disease or fibrosis
3. Development of hematological or solid organ malignancy
4. Presence of an immunodeficiency or abnormal lab values (immunoglobulin or lymphocyte profile)
5. Presence of an endocrine disorder or abnormal hormonal levels
6. Presence of a vascular abnormality
7. Presence of an abnormal ECG or ECHO. Incidence of IHD over time
8. Presence, development of or rate of progression of cytopenias,lung disease, and liver disease compared between TBD causing mutations
9. Presence of TBD mutation in a family member and its association with cytopenias, short telomeres, and evidence of lung or liver involvement. Presence, development of or rate of progression of cytopenias, lung disease, and liver disease compared between family members with the same mutation
10. Genomic analysis using whole exome sequencing or whole genome sequencing to look for potentially disease causing variants in subjects who meet the clinical phenotype for TBD but do not have a known mutation

Cohort 4 (IBMF):

1. Overall survival
2. Treatment response
3. Development of hematological or solid organ malignancy
4. New medical diagnosis and its relationship to any treatment received
5. Record PNH incidence in IBMF as defined by a clone size of >1% in granulocytes
6. Determine the incidence of iron overload, its course with any IBMF treatments, and its response to chelation therapy
7. Record the outcomes of pregnant subjects
8. The presence of viral and bacterial infections and correlation to worsening cytopenias. Presence of worsening cytopenias after vaccination
9. Presence of IBMF mutation in a family member and its association with cytopenias, and other clinical phenotypes
10. Genomic analysis using whole exome sequencing or whole genome sequencing to look for potentially disease causing variants in subjects who meet the clinical phenotype for TBD but do not have a known mutation

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria. Subjects and their family members who undergo screening but ultimately do not meet criteria for cohorts 1-5 will be removed from the study. Subjects may forgo screening and sign directly onto cohorts 1-5 if they meet criteria based on either prior NIH testing or external examinations. Family members will only be asked to be screened for participation onto this study after confirmation of eligibility by an affected participant.

Cohorts 1-4

* Age >=2 years
* Diagnosis of acquired or inherited bone marrow failure or ineffective hematopoiesis or TBD (see below for cohort 3 specific criteria)
* Ability and willingness to come to the NIH CC for consultation and testing
* Ability of subject or Legally Authorized Representative (LAR) to understand the investigational nature of the protocol and their willingness to sign a written informed consent document.
* For cohort 3 - TBD:

Presence of a pathogenic, likely pathogenic, or known family mutation in a telomere maintenance gene

OR

If mutation negative or VUS, telomere length <10th percentile in lymphocytes with at least two clinical features: 1) cytopenia (Hb <10g/dL or ANC <1.5x10^9 or platelets <100), 2) documented liver fibrosis by histology OR abnormal liver US / fibro scan consistent with fatty liver or fibrosis), 3) documented pulmonary fibrosis by histology / radiology OR PFTs showing FEV1 <80% or DLCO <60%, 4) family history of: marrow failure, myeloid malignancy, liver fibrosis or lung fibrosis.

Cohort 5

* Age >= 2 years
* First degree family member with a known or suspected inherited bone marrow failure syndrome from a patient enrolled on this or another NIH protocol as determined by a PI or AI
* Ability and willingness to safely provide blood, buccal swab, or fibroblasts for testing as stated by subject
* Ability of subject or Legally Authorized Representative (LAR) to understand the investigational nature of the protocol and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

-None

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Severe Aplastic Anemia, other acquired marrow failure syndromes, and inherited marrow failure syndromes. Family members of subjects with either suspected or confirmed inherited bone marrow failure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2041-02-04 (Estimated); Study Completion 2041-02-04 (Estimated)

PRIMARY OUTCOMES:
Cohort 4: Rate of progression to transfusion dependent marrow failure, marrow failure requiring therapeutic intervention (such as medical therapy or HSCT) or the progression to hematological malignancy | 20 years
  Rate of progression to transfusion dependent marrow failure, marrow failure requiring therapeutic intervention (such as medical therapy or HSCT) or the progression to hematological malignancy.
Cohort 3: Development of cytopenias, lung disease or liver disease, or (if present at baseline) characterization, and rate of progression of cytopenias, lung disease or liver disease in TBD patients and looking at their overall contribution to m... | 20 years
  Development of cytopenias, lung disease or liver disease, or (if present at baseline) characterization, and rate of progression of cytopenias, lung disease or liver disease in TBD patients and looking at their overall contribution to morbidity and mortality.
Cohort 1: Rate of relapse and clonal evolution in previously treated patients | 20 years
  Rate of relapse and clonal evolution in previously treated patients
Cohort 2: Rate of progression requiring therapeutic intervention | 20 years
  Rate of progression (cytopenias or clonal evolution) requiring therapeutic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Groarke, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a new requirement and the team has yet to discuss the sharing of IPD.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000387-H.html